CLINICAL TRIAL: NCT03388736
Title: Effects of Lavender Oil at Different Concentrations in the Preoperative Waiting Room on Anxiety Levels of Patients Before Orthognathic Surgery
Brief Title: Anxiolytic Effect of Lavender Oil on Orthognathic Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Poyzan Bozkurt, Specialist, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15/10
Record Dates: First submitted 2017-12-08; First posted 2018-01-03 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Anxiety; Osteotomy
Keywords: preoperative; anxiety; orthognathic surgery; lavender oil
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No lavender (No Intervention): No mist will be diffused into the environment.
- 0,1 lavender (Active Comparator): 0,1 ml lavender oil diluted in 120 ml water will be diffused into the environment with (17-33 ml mist output per hour).
  Interventions: Behavioral: Supplementary Medicine
- 0,3 lavender (Active Comparator): 0,3 ml lavender oil diluted in 120 ml water will be diffused into the environment with (17-33 ml mist output per hour).
  Interventions: Behavioral: Supplementary Medicine

INTERVENTIONS:
Behavioral: Supplementary Medicine — A diffuser containing 120 ml water and 0.1 or 0.3 ml lavender oil (according to arm) will be set into the patients' rooms to mist at least 30 minutes before the patients arrive.
  Arms: 0,1 lavender; 0,3 lavender

SUMMARY:
The aim of this study is to determine the possible reducing effects of different concentrations of lavender oil on preoperative anxiety in orthognathic surgery patients who have high anxiety during preoperative wait.

DETAILED DESCRIPTION:
Preoperative anxiety is a common problem. It has long been known that surgical operations, unconsciousness, the risks of the operation itself, and the pain to be encountered in the future can cause a considerable amount of anxiety. Anxiety is associated with an uncertain psychological distress, and may vary to minor disturbances to extreme stress. Depending on the severity of the anxiety, preoperative anxiety can affect how well the patient understands the information about the surgery. In addition, stress factors such as interleukins released in the body in anxiety may negatively affect both surgical and post-surgical periods. We want to help patients improve their satisfaction by reducing their anxiety levels and ensure they have a better surgical experience. In addition, anxiety can also prevent active participation in the treatment of the patient during postoperative recovery. Sedatives and other anxiolytic agents may be prescribed to prevent this condition. However, these methods can have side effects. The physical and psychological effects of essential oils and traditional medicine practices as aromatherapy has been used for a long time and has potency to reduce using sedatives. Lavender oil is a fragrance that many of us have experienced in growing up at home and is also popular today. The lavender plant belongs to the Labitae family and has been used for centuries in dried or essential oil form. Lavender obtained from flower heads and leaves with vapor distillation. Traditionally, this oil is believed to be beneficial for antibacterial, antifungal, muscle relaxant, sedative, antidepressant effects and for burn and insect bites. Nowadays it is used for aromatherapy and antibacterial and pleasant fragrance material which is used in soaps and cosmetic products. This oil has also been specifically investigated and is an essential oil scientifically shown to reduce patient anxiety before various surgeries. However, the anxiolytic effect of this essential oil has not been investigated for orthognatic surgery patients and there is very few studies investigating different concentrations.

The aim of our study is to investigate whether the different concentration of lavender oil diffused in the preoperative environment of orthognathic surgery patients reduces preoperative anxiety.

ELIGIBILITY:
Inclusion Criteria:

* To undergo orthognathic surgery
* To be over 18 years old.
* Volunteering to fill pre-operative anxiety tests

Exclusion Criteria:

* Hypersensitivity to lavender and its products.
* Being on any medication.
* Being a psychiatric or psychological problem and being under treatment.
* Current upper airway infection or asthma story.
* Not want to be involved in the work.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Reduction of preoperative anxiety | STAI will be applied at administration and after 1 hour waiting time.
  State Trait Anxiety Inventory (STAI) questionnaire will be applied. Turkish STAI consists of 2 questionnaires. The first survey measures state anxiety, while the second survey measures continuing anxiety.The State and Trait Anxiety Inventory-STAI (State and Trait Anxiety Scale) is a self-assessing and self-reporting anxiety questionnaire. The reliability and validity of the questionnaire are proven by numerous studies and the Turkish version is a reliable and valid questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Poyzan Bozkurt, DDS PhD, Study Director — Ankara University Faculty of Dentistry
Locations (1):
- Ankara University Faculty of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No